CLINICAL TRIAL: NCT05430984
Title: Outcomes of Mesh Fixation Versus Non Fixation in Laparoscopic TAPP Inguinal Hernia Repair; A Randomized Controlled Clinical Trial
Brief Title: Outcomes of Mesh Fixation Versus Non Fixation in Laparoscopic TAPP Inguinal Hernia Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Ahmed Aouf, Dr, assistant lecturer of General Surgery, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MKSU50-6-16
Record Dates: First submitted 2022-06-20; First posted 2022-06-24 (Actual); Last update posted 2022-06-24 (Actual); Status verified 2022-06

CONDITIONS: Hernia, Inguinal
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laparoscopic TAPP inguinal hernia repair with mesh fixation (Active Comparator): the mesh will be fixed to the abdominal wall using suture, spiral tacks.
  Interventions: Procedure: Laparoscopic TAPP inguinal hernia repair
- Laparoscopic TAPP inguinal hernia repair without mesh fixation (Active Comparator): the mesh will be left as it is and the operation will be concluded
  Interventions: Procedure: Laparoscopic TAPP inguinal hernia repair

INTERVENTIONS:
Procedure: Laparoscopic TAPP inguinal hernia repair — Isolation of preperitoneal space will be accomplished to guarantee the mesh flattening with the medial border at the pubic symphysis, the lateral border at the psoas major and anterior superior iliac spine, superior border at least 3 cm above the conjoined tendon, medial inferior border 3 cm below the pectineal ligament, and lateral inferior border to permit perietalization of the spermatic cord (6-8 cm isolation of the hernia sac and spermatic cord).
  For the mesh fixation group, the mesh will be fixed to the abdominal wall using suture, spiral tacks, whereas for the non-fixation group it will be left as it is and the operation will be concluded. A mesh measuring 15x10cm is placed in the preperitoneal space and fixed using limited numbers of tacks or suture. In some cases, based on body habitus, a slightly smaller mesh could be used. The peritoneum will be closed over the mesh.

SUMMARY:
This work aims to study the outcomes of mesh fixation versus non-fixation of laparoscopic TAPP inguinal hernia repair as regards postoperative pain, recurrence, operative time, and other postoperative complications.

DETAILED DESCRIPTION:
This is a randomized controlled clinical trial that will be conducted on patients who will undergo laparoscopic TAPP inguinal hernia repair in the General Surgery Department. Adult patients of either gender, aged between 18 and 65 years, who had early diagnosed inguinal hernia (unilateral or bilateral) were included. We excluded patients with a recurrent hernia, inguinoscrotal hernia, complicated hernia (incarcerated or strangulated), known ascites or connective tissue disease, heart and kidney failure, and hypoalbuminemia.

Surgery will be performed under general anaesthesia with endotracheal intubation. Patients will be placed in the Trendelenburg position with access to the abdominal cavity through the umbilical port; then, pneumoperitoneum is obtained at 15 mmHg. After pneumoperitoneum, a laparoscope will be inserted through the umbilical incision. The second and third holes will be made on the abdominal median line's left and right side at the umbilical level.

When entering the abdominal cavity, the peritoneum will be cut open in a curved shape 3 cm to the superior margin of the defect. To avoid urinary bladder injury, the medial border of the incision won't cross the medial umbilical ligament. Special attention will be paid to avoid inferior epigastric artery injury while cutting open the peritoneum in the medial part.

When the sac of the oblique hernia enters the internal ring, it will be isolated as much as possible. If there is a large lipoma outside the hernia sac will also be excised. Isolation of preperitoneal space will be accomplished to guarantee the mesh flattening with the medial border at the pubic symphysis, the lateral border at the psoas major and anterior superior iliac spine, superior border at least 3 cm above the conjoined tendon, medial inferior border 3 cm below the pectineal ligament, and lateral inferior border to permit perietalization of the spermatic cord (6-8 cm isolation of the hernia sac and spermatic cord). The patient is tilted head-down position.

For the mesh fixation group, the mesh will be fixed to the abdominal wall using suture, spiral tacks, whereas for the non-fixation group it will be left as it is and the operation will be concluded. A mesh measuring 15x10cm is placed in the preperitoneal space and fixed using limited numbers of tacks or suture. In some cases, based on body habitus, a slightly smaller mesh could be used. The peritoneum will be closed over the mesh to reduce the risk of mesh adhesion to intestines, erosion, fistula formation, and small bowel obstruction by one of three methods: suture, or tack closure.

Operative data will be collected as regard operative time, the effect on chronic pain and quality of life, recurrence, and other complications (seroma, urine retention)

ELIGIBILITY:
Inclusion Criteria:

* Adult patients of either gender, aged between 18 and 65 years, who had early diagnosed inguinal hernia (unilateral or bilateral)

Exclusion Criteria:

* patients with a recurrent hernia, inguinoscrotal hernia, complicated hernia (incarcerated or strangulated), known ascites or connective tissue disease, heart and kidney failure, and hypoalbuminemia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
postoperative pain | 12 months
  the degree of pain after surgery in the inguinal region assessed by numerical rating score

CONTACTS AND LOCATIONS:
Locations (1):
- Kafrelsheikh University, Kafr ash Shaykh, Kafr el-Sheikh Governorate, Egypt